CLINICAL TRIAL: NCT05319782
Title: Long-term Assesment of Patients Operated for Hypospadias in Their Childhood : Urinary, Aesthetical, Sexual and Psycho-social Consequences
Acronym: SAHARA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021/663
Record Dates: First submitted 2022-04-01; First posted 2022-04-08 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Hypospadias
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental)
  Interventions: Other: Urethral stenosis assesment

INTERVENTIONS:
Other: Urethral stenosis assesment — Auto-questionnaires + Clinical examination + Flow metry and post-mictional residue

SUMMARY:
The purpose of this study is to assess the long term urinary, sexual, cosmetic and psycho-social outcomes of adult patients operated for hypospadias during childhood

ELIGIBILITY:
Inclusion Criteria:

* Patients operated for hypospadias during childhood (before the age of 15) at the University Hospital of Besançon (France)

Exclusion Criteria:

* Patients with a non-operated hypospadias
* Opposition to participate
* Legal incapacity

Ages: 18 Years to 23 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 66 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of adult patients with urethral stenosis following a repair surgery performed during childhood | Day 1
  Proportion of adult patients with urethral stenosis following a repair surgery performed during childhood, assessed with flowmetry (maximal urinary flow)

CONTACTS AND LOCATIONS:
Overall Officials: Yann CHAUSSY, MD, PhD, Principal Investigator — CHU De Besançon
Locations (1):
- CHU de Besançon, Besançon, France